CLINICAL TRIAL: NCT00037557
Title: An Open-Label, Single-Arm, Safety and Efficacy Study of Recombinant Human Factor IX (rFIX; BeneFIX®) in Children Less Than 6 Years of Age With Severe Hemophilia B
Brief Title: Study Evaluating rFIX; BeneFIX in Severe Hemophilia B
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3090A1-301
Record Dates: First submitted 2002-05-17; First posted 2002-05-20 (Estimated); Last update posted 2007-12-27 (Estimated); Status verified 2007-12

CONDITIONS: Hemophilia B
Keywords: Hemophilia B
MeSH Terms: conditions — Hemophilia B | interventions — Factor IX

INTERVENTIONS:
Drug: BeneFIX

SUMMARY:
To characterize the safety and efficacy of rFIX in children less than 6 years of age with severe hemophilia B in the setting of acute bleeding episodes, prophylaxis, and/or surgery.

This study will provide an opportunity for systematic observation of treatment with rFIX in children less than 6 years of age regardless of prior FIX treatment. Younger patients exhibit a different pharmacokinetic profile and therefore may respond differently to rFIX infusions when compared with older children and adults. This evaluation will provide data from which recommendations can be made regarding rFIX dosing and treatment of these patients. Surveillance for certain observations that have been made in patients treated with rFIX in the clinical and postmarketing setting will be performed, including inhibitor development, thrombogenicity, FIX recovery/lack of effect, allergic-type manifestations, and RBC agglutination. Comparisons will be derived from published reports and communications describing experience with other FIX products and protein therapeutics in general.

ELIGIBILITY:
Inclusion Criteria:

* Severe hemophilia B
* Less than 5 years of age
* In the investigator's judgment, the patient and/or caregiver will be compliant to study procedures

Exclusion Criteria:

* A currently detectable FIX inhibitor. A family history of inhibitors will not exclude the patient.
* Impaired liver function
* Impaired renal function

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20
Dates: Start 2002-09; Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
To characterize the safety and efficacy of rFIX in children less than 6 years of age with severe hemophilia B in the setting of acute bleeding episodes, prophylaxis, and/or surgery.

SECONDARY OUTCOMES:
To measure the incremental recovery of rFIX in children following a 75-IU/kg bolus infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, MD, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (6):
- United States (6):
  - Aurora, Colorado
  - Detroit, Michigan
  - New Brunswick, New Jersey
  - Chapel Hill, North Carolina
  - Dayton, Ohio
  - Houston, Texas

REFERENCES:
- [Derived] Wojciechowski J, Gaitonde P, Hughes JH, Ravva P. Population Modeling of Factor IX Activity Following Administration of Fidanacogene Elaparvovec Gene Therapy in Participants with Hemophilia B. Clin Pharmacokinet. 2025 Oct;64(10):1531-1548. doi: 10.1007/s40262-025-01535-y. Epub 2025 Aug 1. PMID 40750723
- [Derived] Rendo P, Smith L, Lee HY, Shafer F. Nonacog alfa: an analysis of safety data from six prospective clinical studies in different patient populations with haemophilia B treated with different therapeutic modalities. Blood Coagul Fibrinolysis. 2015 Dec;26(8):912-8. doi: 10.1097/MBC.0000000000000359. PMID 26196195